CLINICAL TRIAL: NCT05851937
Title: Optimizing Language Outcomes for Young Adults With Intellectual and Developmental Disabilities: A Written Language Intervention Using Functional Texts
Brief Title: Written Language Intervention for Adults With Intellectual and Developmental Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BaylorU; R21DC020787 (NIH)
Record Dates: First submitted 2023-04-14; First posted 2023-05-10 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Intellectual Disability; Developmental Disability
MeSH Terms: conditions — Intellectual Disability; Developmental Disabilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Written language intervention (Experimental): Participants will receive 3 months of weekly written language intervention sessions via telepractice.
  Participants will be assessed at three time points to monitor outcomes.
  Interventions: Behavioral: Written language intervention
- Periodic language check-up (No Intervention): Participants will be assessed at three time points to monitor outcomes.

INTERVENTIONS:
Behavioral: Written language intervention — Young adults with Intellectual and Developmental Disabilities (IDD) are taught reading comprehension strategies in three phases (before, during, after) using a graphic organizer as visual support. At the beginning of each phase, the interventionist: (a) defines the strategies, (b) describes and models how to use the strategies, and (c) answers questions about the strategies. Then the participant practices the strategies during 45-min sessions, two times per week, over 3 months. Each session follows the teach-model-coach-review format, the interventionist: (a) reviews the strategies (5 min), (b) models the strategies using a think-aloud (10 min), (c) prompts the participant to practice the strategies with support (15 min), (d) prompts the participant to use a think-aloud to practice the strategies independently using a functional literacy text (10 min), and (e) reviews and summarizes the session (review; 5 min).
  Arms: Written language intervention

SUMMARY:
The purpose of this study is to evaluate the effects of a written language intervention using functional texts for young adults with intellectual and developmental disabilities.

DETAILED DESCRIPTION:
Individuals with intellectual and developmental disabilities (IDD) often present with limited literacy achievement which results in an absence of opportunities to foster written language development. However, when young adults with IDD are provided opportunities to broaden their literacy education even after high school, they continue to develop and improve their written and spoken language skills, which is associated with improved vocational and independent living options. To date, few studies have examined effective communication interventions for the often-underrepresented population of young adults with IDD. The objective of this study is to examine the feasibility, acceptability, and initial effectiveness of a functional written language intervention embedded in naturally occurring daily activities (e.g., text messages, emails) for young adults with IDD. The central hypothesis is that (a) explicit written language intervention for functional texts (WLIFT) will result in greater use of reading comprehension strategies before, during, and after reading and (b) use of reading comprehension strategies will be associated with improvements in written and spoken language outcomes. The specific aims include (1) examining the effects of WLIFT intervention on use of reading comprehension strategies in functional texts by young adults with IDD, 2) examining the effects of the intervention on distal written language outcomes, and (3) examining the effects of the intervention on distal spoken language outcomes. The study target enrollment includes 40 young adults with IDD who will be randomly assigned to either the treatment or control group. Individuals in both groups will be assessed: (a) at the start of the study, (b) at the conclusion of intervention, and (c) six months following the conclusion of intervention. Individuals with IDD in the WLIFT group will receive 3-months of intervention that: (a) utilizes functional texts-activities of daily living that involve written language (e.g., text messages), (b) is specifically designed based on the phenotype of commonly occurring IDDs and is delivered at a critical time as young adults transition to independence, (c) involves teaching and assessing comprehension strategies implemented before, during, and after reading that have been previously shown to be associated with stronger written and spoken language skills in struggling readers, and (d) is implemented via telepractice to promote service delivery in meaningful contexts for the individual with IDD. This research is significant because it is expected to apply, adapt, and evaluate written language strategies found to be effective in other populations of struggling readers, thereby advancing the field of language development in individuals with IDD, where there is a striking paucity of communication intervention research.

ELIGIBILITY:
Inclusion Criteria:

* intellectual and/or developmental disability
* correctly read at least 80% of words on word reading screener
* have functional literacy needs
* English as primary spoken language and use oral communication as their primary form of communication
* normal or corrected to normal vision

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor University, Waco, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Written Language Intervention: Participants will receive 3 months of weekly written language intervention sessions via telepractice.
  Participants will be assessed at three time points to monitor outcomes.
  Written language intervention: Young adults with Intellectual and Developmental Disabilities (IDD) are taught reading comprehension strategies in three phases (before, during, after) using a graphic organizer as visual support. At the beginning of each phase, the interventionist: (a) defines the strategies, (b) describes and models how to use the strategies, and (c) answers questions about the strategies. Then the participant practices the strategies during 45-min sessions, two times per week, over 3 months. Each session follows the teach-model-coach-review format, the interventionist: (a) reviews the strategies (5 min), (b) models the strategies using a think-aloud (10 min), (c) prompts the participant to practice the strategies with support (15 min), (d) prompts the participant to use a think-aloud to practice the strategies independently using a functional literacy text (10 min), and (e) reviews and summarizes the session (review; 5 min).
Period: Overall Study
Arm/Group | Written Language Intervention | Periodic Language Check-up
Started | 25 | 23
Completed | 23 | 21
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Written Language Intervention | Periodic Language Check-up | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.65 (5.13) | 22.74 (2.49) | 22.17 (4.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 15 | 8 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 19 | 15 | 34
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 23 | 21 | 44
Phonological Awareness Literacy Screening-Kindergarten Word Recognition Subtest [Mean (Standard Deviation); unit: scores on a scale] — The PALS-K: Word Recognition primer is a subtest designed to measure students' ability to recognize and read familiar words, reflecting early word-level reading skills and automaticity.
  The Word Recognition subtest score ranges from 0 to 20, representing the total number of words correctly identified which was then reported as a percentage accuracy score. Higher scores indicate better outcomes, reflecting stronger word recognition skills, while lower scores indicate weaker performance.
  scores on a scale | 97.39 (4.71) | 98.33 (2.42) | 97.84 (3.8)
Woodcock Reading Mastery Tests-III Word Identification [Mean (Standard Deviation); unit: raw score] — The WRMT-III Word Identification subtest measures single-word reading accuracy, specifically the ability to correctly identify and read real printed words.
  The raw score for Word Identification represents the total number of words read correctly. Raw scores range from 0 to 46. Higher raw scores indicate better outcomes, reflecting stronger word recognition skills, while lower scores indicate weaker performance. The Word Identification raw score was reported independently.
  raw score | 26 (6.05) | 27.33 (5.72) | 26.64 (5.86)
Woodcock Reading Mastery Tests-III Word Attack [Mean (Standard Deviation); unit: raw score] — The WRMT-III Word Attack subtest measures phonetic decoding skills, specifically the ability to apply letter-sound relationships to read unfamiliar or nonsense words.
  The raw score for Word Attack represents the total number of nonwords read correctly. Raw scores range from 0 to 26. Higher raw scores indicate better outcomes, reflecting stronger word recognition skills, while lower scores indicate weaker performance. The Word Attack raw score was reported independently.
  raw score | 12.09 (7.12) | 10 (6.31) | 11.09 (6.75)
Woodcock Reading Mastery Tests-III Passage Comprehension [Mean (Standard Deviation); unit: raw score] — The WRMT-III Passage Comprehension subtest assesses reading comprehension, specifically the ability to derive meaning from text using a cloze (fill-in-the-blank) format.
  The raw score for Passage Comprehension represents the total number of nonwords read correctly. Raw scores range from 0 to 38. Higher raw scores indicate better outcomes, reflecting stronger word recognition skills, while lower scores indicate weaker performance. The Passage Comprehension raw score was reported independently.
  raw score | 11.57 (4.89) | 13.95 (5.19) | 12.70 (5.12)
Kaufman Brief Intelligence Test-2 Revised [Mean (Standard Deviation); unit: raw score] — The KBIT-2R is a standardized measure of general intellectual ability that includes Verbal Ability and Nonverbal Ability subscales, which measure verbal reasoning/vocabulary and nonverbal problem solving, respectively.
  Raw scores from the two subscales are combined and converted using age-normed scoring procedures to yield an IQ Composite score. The IQ Composite is reported on a standard score scale with a mean of 100 and a sd of 15, with scores ranging approximately from 40 to 160. Higher scores indicate better cognitive performance, while lower scores indicate weaker performance.
  raw score | 60.48 (10.32) | 63.9 (12.04) | 62.11 (11.18)

OUTCOME MEASURES:

1. Primary Outcome: Use of Reading Comprehension Strategies
Description: Total number of different reading comprehension strategies used correctly. A blank version of the FRAME intervention graphic organizer including only the picture icons of the reading comprehension strategies was displayed alongside a functional text stimulus (e.g., text messages, e-mails) that was designed to closely reflect participants' daily written communications. the examiner prompted the participant to begin reading the functional text. Each think-aloud was scored for the participants' accurate use of reading comprehension strategies. A percent accuracy score was calculated based on (a) the total number of strategies implemented correctly (out of nine; excluding Strategy 4 [read text aloud] because all participants were expected to read the text) and (b) implementing the strategies at the appropriate time (before, during, after reading) to earn up to three additional points (max score = 12). Higher scores reflect better performance.
Time Frame: 3 months after start of intervention
Measure: Mean (Standard Deviation); unit: reading comprehension strategies used
Arm/Group | Written Language Intervention | Periodic Language Check-up
Number analyzed (Participants) | 23 | 21
reading comprehension strategies used | 3.986 (5.019) | 0.032 (.256)

2. Secondary Outcome: Reading Comprehension of Functional Texts
Description: Percentage of multiple choice comprehension questions answered correctly. The interventionist prompted the participant to read a functional text stimulus aloud and then prompted the participant to answer five (two literal, three inferential) multiple-choice questions that were read aloud by the interventionist. This task was repeated across a total of six functional literacy stimuli, two in each of the following domains-employment, independent living, and social. A percent accuracy score was calculated for each of the functional literacy stimuli, and a total average score was reported across all functional literacy stimuli. Higher scores reflect better performance.
Time Frame: 3 months after start of intervention
Measure: Mean (Standard Deviation); unit: proportion of questions
Arm/Group | Written Language Intervention | Periodic Language Check-up
Number analyzed (Participants) | 23 | 21
proportion of questions | .572 (.613) | .127 (.505)

3. Secondary Outcome: Use of Spoken Language to Indicate Comprehension
Description: Respond to functional text using spoken modality. The assessor displayed a functional text and prompted the participant to help them verbally respond to the functional text sample. All the functional texts utilized in the spoken language measure requested three pieces of information (e.g., state your name, e-mail, T-shirt size) and thus were scored using a 4-point (0-3) rubric rating with 1 point awarded for each piece of information provided. Higher scores reflect better performance. This task was repeated across a total of six functional literacy stimuli, two in each domain; an average score was reported.
Time Frame: 3 months after start of intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Written Language Intervention | Periodic Language Check-up
Number analyzed (Participants) | 23 | 21
score on a scale | .051 (.704) | .333 (.643)

4. Secondary Outcome: Spoken Language: Summarize
Description: Verbal summary of functional text. The assessor displayed a functional text and prompted the participant to read the text and then provide a summary of all the important information. Summaries were scored using a rubric that evaluated content, accuracy, paraphrasing, and organization each using a 4-point (0-3) scale. Higher scores reflect higher performance.
Time Frame: 3 months after start of intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Written Language Intervention | Periodic Language Check-up
Number analyzed (Participants) | 23 | 21
score on a scale | .780 (1.302) | .217 (1.119)

ADVERSE EVENTS:
Time Frame: through study completion, an average of 9 months
Arm/Group | Written Language Intervention | Periodic Language Check-up
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21
Other Adverse Events (participants affected / at risk) | 0/23 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT05851937/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT05851937/ICF_002.pdf